CLINICAL TRIAL: NCT06786598
Title: The Effect of Body Mass Index and Total Cholesterol Levels on Histopathological Grading in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Breast cancer grading; Institutional review board (Other: Tishreen university)
Record Dates: First submitted 2025-01-12; First posted 2025-01-22 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cholesterol titration (Experimental)
  Interventions: Diagnostic Test: Cholesterol

INTERVENTIONS:
Diagnostic Test: Cholesterol — Qimica/kit

SUMMARY:
Breast cancer is a widespread cancer that affects high percentiles of women worldwide.The development and aggressiveness of breast cancer cells can be evaluated depending on the histopathological grading which reflects the degree of differentiation. Several factors related to lifestyle can impact the development of breast cancer. Obesity is an important factor that received the attention in recent years. The using of body mass index(BMI) is still the common method for identifying obesity which is defined when having 30kg/m² or more. Previous epidemiological and clinical studies found that obesity was correlated with advanced breast cancer especially in postmenopausal patients . Also, the changes in cholesterol levels can influence breast cancer risk in the context of obesity. The findings of other studies is still controversial; many studies revealed that elevated total cholesterol levels could increase breast cancer risk while others found to have no effect. Due to the possibility of previous factors' effect on breast cancer progression, we purposed in this study to assess the association of BMI and total cholesterol with histopathological grading according to menopausal status among a group of breast cancer patients in Syria

ELIGIBILITY:
Inclusion Criteria:

all participants after ensurement that all their clinical and demoghraphical data are completed

Exclusion Criteria:

metabolic syndromes, as well as patients with statin therapy and hormonal replacement treatment.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 85 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Evaluating The effect of body mass index and total cholesterol levels on histopathological grading in breast cancer patients | baseline
Assessing the body mass index between patients via dividing weight(in killogram) by height (in meter squared) | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Tishreen university, Latakia, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Llaverias G, Danilo C, Mercier I, Daumer K, Capozza F, Williams TM, Sotgia F, Lisanti MP, Frank PG. Role of cholesterol in the development and progression of breast cancer. Am J Pathol. 2011 Jan;178(1):402-12. doi: 10.1016/j.ajpath.2010.11.005. Epub 2010 Dec 23. PMID 21224077